CLINICAL TRIAL: NCT05152745
Title: Effect of Ginger Extract on Postprandial Glycemia of Healthy Adults and Its Antioxidant Properties: a Randomized Controlled Trial
Brief Title: Effect of Ginger Extract on Postprandial Glycaemia of Healthy Adults and Its Antioxidant Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 519ginger
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Hyperglycemia, Postprandial
Keywords: Ginger, hyperglycemia, antioxidant, phenols, flavonoids
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (OGTT) (Placebo Comparator): The control group participants ingested glucose solution alone (OGTT) prepared with 75 g of anhydrous oral glucose as prescribed by the ADA, dissolved in 200 ml of water.
  Interventions: Other: Placebo OGGT
- Intervention (OGTT plus Ginger extract) (Experimental): The intervention group ingested glucose solution followed by 100 ml of ginger aqueous extract (0.2g ginger, each dose).
  Interventions: Other: Ginger aqueous extract

INTERVENTIONS:
Other: Placebo OGGT — After overnight fasting, blood glucose level was assessed through a capillary drop blood The control group participants ingested glucose solution alone (OGTT) prepared with 75 g of anhydrous oral glucose as prescribed by the ADA, dissolved in 200 ml of water. Blood glucose level was also measured at 30 (t30), 60 (t60), 90 (t90) and 120 (t120) minutes immediately after intervention, for each participant, in control and intervention groups.
  Glucometer equipment, strips for glucose meters (One Touch Select Plus) and sterilized lancets (Sarstedt normal 21G) were used to measure blood glucose concentrations, taking due care of safety and asepsis.
  Arms: Placebo (OGTT)
Other: Ginger aqueous extract — After overnight fasting, blood glucose level was assessed through a capillary drop blood The intervention group participants ingested glucose solution alone (OGTT) prepared with 75 g of anhydrous oral glucose as prescribed by the ADA, dissolved in 200 ml of water, followed by 100mL of ginger extract (0.2g). Blood glucose level was also measured at 30 (t30), 60 (t60), 90 (t90) and 120 (t120) minutes immediately after intervention, for each participant, in control and intervention groups.
  Glucometer equipment, strips for glucose meters (One Touch Select Plus) and sterilized lancets (Sarstedt normal 21G) were used to measure blood glucose concentrations, taking due care of safety and asepsis.
  Arms: Intervention (OGTT plus Ginger extract)

SUMMARY:
Background: Hyperglycemia is a risk factor to disease development, namely, diabetes mellitus. The blood glucose level management, particularly on post-prandial period has an important role in the prevention of different diseases. Ginger is a specie that has been demonstrated a benefit effect on glycaemia on diabetes.

Aim: The aim of this study was 1) to investigate the effects of ginger infusion in the glycaemic response in nondiabetic adults; 2) to evaluate total phenolic content the antioxidant activity of Ginger (Zingiber officinale Roscoe) aqueous extracts.

Methodology: 24 nondiabetic subjects were randomly allocated into two groups: intervention group (GI; n=15) and control group (GC; n=15). An oral glucose solution (OGTT) and an OGTT following ginger extract solution were administrated in control and intervention groups, respectively. Blood glucose levels were measurement at fasting and after 30, 60, 90 and 120 minutes after interventions in both groups. Total phenolic content and flavonoids compounds determination of the aqueous ginger extract was determined according to Prabha method. Antioxidant activity was also measured through ABTS method and free radicals inhibition capacity. Repeated Measures ANOVA of mixed type and independent samples t-test were used in statistical analysis.

DETAILED DESCRIPTION:
This clinical trial was approved by Ethical Committee (process number 519 at 23 November 2016). All participants signed a written informed consent after aim and experimental risk procedures explanation and its protected confidentiality was guaranteed. The experimental procedure involving human was care out according Declaration of Helsinki.

This blind (to participants) randomized controlled clinical trial was conducted at Egas Moniz higher education school in 30 nondiabetic adults. Participants with ages between 18 and 40 were selected and randomly allocated in intervention group (IG) (n=15) and control group (CG) (n=15), in which participants were alternated include in the groups. The IG performed an oral glucose tolerance test (OGTT) followed by aqueous ginger extract administration and the CG performed an OGTT administration alone.

For ginger extract preparation, powder ginger (Zingibre officinalle Roscoe) was obtained from Portugal Company with India origin and stored in a dried environmental locally until needed. The product has a batch number of LI1GIGRNT150012. Powder ginger was individually weight (0.2g each dose) and added to 100mL of boiled water obtaining the ginger extract, infusing 10 minutes. Ginger extract solution was after cooled at room temperature and distributed to each participant. This method was adapted by Wilkinson, J. M. (2000). For chemical analysis, a aqueous ginger extract previously obtained was used.

Regarding to blood glucose level assessment, the blood sample were collected for each participant using a capillary drop blood before the intervention (fasting) and after 30, 60, 90 and 120 minutes. The blood glucose level analysis was performed using a strips for glucose meter (Onetouch Select Plus Flex), a sterilized lancet and a glucose meter equipment.

General characteristics data of the participants were collected, namely, anthropometrics data, pharmacologic treatment and medical condition using a questionnaire. In addition, a 24-hour dietary recall at the day before the intervention was employing to sample participants. The nutritional analyzed of diet ingested was performed by Food Processor SQL (version 10.5.0).

The total phenolic compounds determination of the aqueous ginger extract was determined according to Folin-Ciocalteu method. The total phenolic results were expressed as mg gallic acid equivalent (GAE)/L of ginger extract. A volume of 125 μL of ginger extract and 2 mL of sodium carbonate were added to 2.5 mL of Folin-Ciocalteu reagent. After 15 min the absorbance was measured at 765 nm. The flavonoids compounds determination of the aqueous ginger extract was determined according to Prabha method. The flavonoids results were expressed as mg quercetin equivalent (GAE)/L of ginger extract. A volume of 2 mL of ginger extract were added to 0.1 mL of aluminum chloride anhydrous solution (10%), 0.1 mL of potassium acetate (1M) and 2.8 mL of distilled water. After 30 min the absorbance was measured at 415 nm.

The antioxidant activity was measured through different assays:

The superoxide anion radicals scavenging activity was determined based on Morais et al method. Superoxide anion was generated by reacting phenazine methosulfate (PMS), nicotinamide adenine dinucleotide hydride (NADH), and oxygen causing reduced NBT in Formazan. A volume of 0.5mL of sample was added to 0.5mL of a solution containing NADH (189 microM) and NBT (120 microM) with Tris-HCl (40mM, pH = 8). The reaction started after the addition of 0.5mL of PMS (60microM). Control sample was measured using only distilled water. After 5min of incubation, control absorbance was measured at 560 nm at room temperature.

The nitric oxide inhibitory activity was determined according Khayami et al method. A volume of 1mL of sodium nitroprusside 10nm was added to 250microL de phosphate buffered saline (PBS) and 250microL of test solution and it was shaken. The previous solution was incubated for 150 min at 25ºC and following add 3mL of sulfanilic acid and 0.33% of acetic acid glacial. After 5 min at room temperature, it was add 3mL of n-(1-naphthyl)ethylenediamine dihydrochloride (NED, 0.1% m/v) and incubated for 30 min at 25ºC. The absorbance was measured at 533nm. The previous procedure was employed to control obtained using water.

The free radical 2,2'-azino-bis (3-ethylbenzothiazoline-6-sulfonic acid) (ABTS) was obtained by ABTS oxidation with potassium persulfate 140mM for 12h in dark, according Zulueta et al method. It was prepared a solution with 10mL ABTS 7nm and 176microL persulfate and storage at room temperature by 12h in dark. The previous solution was diluted with ethanol until 0.7 absorbance at 734nm. A volume of 2850microL of ABTS radical was added to 150microL of sample and to 150microL of water. After 30min in dark the absorbance was determined at 734nm. The Trolox concentration was using as standard (mM Trolox/L). This test was performed for several extract concentrations in order to calculate IC50.

Data statistical analysis was performed using SPSS Statistics (Statistical Package for Social Sciences) (version 22) software. Mean and standard error of the mean were used. Shapiro-Wilk and Repeated Measures ANOVA of mixed type were used. Independent samples T-test was used to assess the difference between the 2 groups for total caloric value, carbohydrates, protein and lipid ingested, Cmax (maximum concentration), ΔCmax (variation of maximum concentration), and AUC (area under the curve) Incremental values. The AUC was calculated by Software GraphPad Prim (version 7.03). All statistical tests were performed at the 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* subjects without glucose metabolism alteration

Exclusion Criteria:

* medication for glycemia
* had gastrointestinal symptoms or disease
* pregnancy or lactation
* had allergy to ginger.
* to ingest ginger at the day before the intervention.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose levels time curve | up to 120 minutes after intervention
  Mean blood glucose levels (mmol/L) obtained after oral glucose tolerance test in control group and after oral glucose tolerance test plus baobab extract in intervention group at different moments
Incremental area under the curve of glucose levels | At 120 minutes after intervention
  the blood glucose incremental area under the curve (AUCi) of each participant was defined using the GraphPad Prism program (version 5.0).
Blood glucose maximum concentrations | At 60 minutos after intervention
  Mean blood glucose levels (mmol/L)
Antioxidant activity determination of Ginger extract | At baseline
  Mean values of anion and radical inhibition capacity and mean values of antioxidant capacity by ABTS (micromol TE/g)
Total phenolic compounds | At baseline
  Mean values of total phenolic compounds (mg of gallic acid/g ginger)
Flavonoids | At baseline
  Mean values of flavonoids (mg quercetin of/g ginger)

SECONDARY OUTCOMES:
Weight of participants | At baseline
  Mean values of weight (in kilograms)
Body mass index of participants | At baseline
  Mean values of body mass index (Kg/m2), calculated as weight (Kg) divided by height (m2) squared (Kg/m2)
Height of participants | At baseline
  Mean values of height (in meters)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernanda Mesquita, Principal Investigator — Centro de Investigação Interdisciplinar Egas Moniz, Instituto Universitário Egas Moniz, Portugal
Locations (1):
- Instituto Universitário Egas Moniz, Almada, Monte de Caparica, Portugal